CLINICAL TRIAL: NCT00988585
Title: Evaluation of the Safety and Biologic Effects of an Eicosapentaenoic (EPA)-Enriched Oil
Acronym: EPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cardiovascular Research Associates (Network)
Collaborators: Dupont Applied Biosciences (Industry)
Responsible Party: Michael Dansinger, MD, Cardiovascular Research Associates
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dupont-0609
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Heart Disease
Keywords: Heart Disease Risk Reduction
MeSH Terms: conditions — Heart Diseases | interventions — Fish Oils; Olive Oil; Oleic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Olive Oil (Placebo Comparator): Olive Oil 600 mg/day
  Interventions: Dietary Supplement: Olive Oil
- EPA 1800 (Active Comparator): 1800 mg/day
  Interventions: Dietary Supplement: EPA 1800
- DHA (Active Comparator): DHA 600 mg/day
  Interventions: Dietary Supplement: DHA
- EPA 600 (Active Comparator): EPA 600 mg/day
  Interventions: Dietary Supplement: EPA 600

INTERVENTIONS:
Dietary Supplement: EPA 600 — EPA 600 mg/day for 6 weeks
  Other Names: omega 3 fat; fish oil
  Arms: EPA 600
Dietary Supplement: EPA 1800 — 1800 mg/day for 6 weeks
  Other Names: omega 3 fat; fish oil
  Arms: EPA 1800
Dietary Supplement: Olive Oil — 600 mg/day for 6 weeks
  Other Names: Oleic acid
  Arms: Olive Oil
Dietary Supplement: DHA — 600 mg/day for 6 weeks
  Other Names: omega 3 fat; fish oil
  Arms: DHA

SUMMARY:
The goal is to test the safety and efficacy of an EPA-enriched oil made by DuPont. DuPont wishes to corroborate the safety of its novel oil rich in EPA in humans prior to placing such a dietary supplement on the market. The goal of this study is to test this oil at doses of 600 mg and 1800 mg of EPA/day as compared to olive oil placebo and a comparator oil providing 600 mg of DHA/day over a 6 wk period. In a parallel arm study design, 120 healthy adults will be randomized to one of four groups (30 in each group) and studied in both the fasting and post-prandial state.

DETAILED DESCRIPTION:
The safety profile of omega-3 fatty acids is considered to be excellent, and has been recognized as safe (GRAS) by the US Food and Drug Administration when EPA and DHA (docosahexanoic acid) are given together at a dose of 3 grams/day or less. Safety will be monitored by assessing for adverse reactions, measuring vital signs and a variety of laboratory tests including a complete metabolic profile and complete blood count. Efficacy will be assessed by measuring changes in fatty acid profile and or fatty acid ratios.

The goal of this study is to test this EPA oil at doses of 600 mg and 1800 mg of EPA/day as compared to olive oil placebo and a comparator oil providing 600 mg of DHA/day over a 6 wk period. In a parallel arm study design, 120 healthy adults will be randomized to one of four groups (30 in each group) and studied in both the fasting and post-prandial state.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or surgically sterile females between ages 21-70.
* BMI of 20-35.

Exclusion Criteria:

* competitive exerciser.
* current smokers.
* those already taking dietary supplements (EPA, DHA, flax seed oil, fish oil, cod liver oil, weight control products, or high doses of vitamin C (> 500 mg/day) or vitamin E (> 400 units/day).
* those consuming more than 3 oily fish species/week.
* those consuming > 2 drinks/day.
* those with a history of a bleeding disorder, or history of significant cardiac, renal, hepatic, gastro-intestinal, pulmonary, neoplastic, biliary or endocrine disorders such as uncontrolled thyroid disease, or uncontrolled hypertension or diabetes.
* those taking medications affecting serum lipids, body weight, or blood clotting.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
No change in safety laboratory tests including comprehensive metabolic profile and complete blood count. | 6 weeks

SECONDARY OUTCOMES:
Efficacy will be assessed by measuring changes in fatty acid profile and or fatty acid ratios. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Dansiner, M.D., Principal Investigator — Cardiovascular Research Associates
Locations (1):
- Cardiovascular Research Associates, Boston, Massachusetts, United States